CLINICAL TRIAL: NCT03922568
Title: Effect of Sperm Selection Techniques on Human Neonatal Gender Ratio in Patients Undergoing ICSI
Status: Completed | Type: Observational
Sponsor: Ganin Fertility Center (Other)
Collaborators: The Cleveland Clinic (Other); University of the Western Cape (Other)
Responsible Party: Principal Investigator, khaled Elqusi, Senior clinical embryologist, Ganin Fertility Center
Other Study IDs: GFC - 003
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Gender Ratio of ICSI Outcome
Keywords: Gender Ratio; PICSI; MACS; Sperm Selection
MeSH Terms: interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Density Gradient Centrifugation (DGC): semen was layered over 50 % and 90% discontinuous Density Gradient layers in a 15ml conical tube, then centrifuged at 250 g for 8 min at room temperature. supernatant was aspirated and the resulted pellet was washed using Sperm wash media and centrifuged at 250 g for 8 min at room temperature. The final pellet was re suspended in residual volume
  Interventions: Other: Density Gradient Centrifugation
- Physiological ICSI (PICSI): Semen processing is done by double layer DGC method followed by adding Sperm to the dot of hyaluronan on the PICSI dish, within minutes the bound sperm are attached by their acrosome to the surface of the dot. Hyaluronan bound sperms are selected for oocyte injection
  Interventions: Device: Physiological ICSI
- Magnetic Activated Cell Sorting (MACS): Semen processing is done by double layer DGC method. The resulted pellet is labeled with Annexin V microbeads followed by separation on MACS column, the eluted fraction contains non apoptotic sperms suitable for oocyte injection.
  Interventions: Device: Magnetic Activated Cell Sorting

INTERVENTIONS:
Other: Density Gradient Centrifugation — semen was layered over 50 % and 90% discontinuous Density Gradient layers in a 15ml conical tube, then centrifuged at 250 g for 8 min at room temperature. supernatant was aspirated and the resulted pellet was washed using Sperm wash media and centrifuged at 250 g for 8 min at room temperature. The final pellet was re suspended in residual volume
  Other Names: DGC
  Groups: Density Gradient Centrifugation (DGC)
Device: Physiological ICSI — Semen processing is done by double layer density gradient method followed by adding Sperm to the dot of hyaluronan on the PICSI dish, within minutes the bound sperm are attached by their acrosome to the surface of the dot. Hyaluronan bound sperms are selected for oocyte injection
  Other Names: PICSI
  Groups: Physiological ICSI (PICSI)
Device: Magnetic Activated Cell Sorting — Semen processing is done by double layer density gradient method. The resulted pellet is labeled with Annexin V microbeads followed by separation on MACS column, the eluted fraction contains non apoptotic sperms suitable for oocyte injection.
  Other Names: MACS
  Groups: Magnetic Activated Cell Sorting (MACS)

SUMMARY:
babies of known gender born out of 388 ICSI cycles were investigated for the gender ratio and then divided into three groups according to the sperm selection technique used before performing sperm injection. Statistical analysis were made to compare ratios and compare results of three arms

DETAILED DESCRIPTION:
A total of 529 babies of known gender born out of 388 ICSI cycles between August 2016 and May 2018 at Ganin Fertility Center, Cairo, Egypt, were investigated for the gender ratio and then divided into three groups according to the sperm selection technique used before performing sperm injection; DGC (237 neonates out of 173 ICSI cycles), PICSI (147 neonates out of 109 ICSI cycles) , and MACS (145 neonates out of 106 ICSI cycles). In PICSI and MACS groups. Power analysis was done by comparing the sex ratio of the neonates between DGC, PICSI and MACS. The chi-squared test for independent samples was chosen to perform the power analysis with α-error level at 0.05. P values less than 0.05 were considered statistically significant. All statistical calculations were done using IBM SPSS (Statistical Package for the Social Science; IBM Corp, Armonk, NY, USA) release 22 for Microsoft Windows.

ELIGIBILITY:
Inclusion Criteria:

* Full Term Delivery
* ICSI cases using DGC for sperm selection
* ICSI cases using MACS for sperm selection
* ICSI cases using PICSI dishes for sperm selection
* Fresh blastocyst stage embryo transfer at
* Fresh ejaculate

Exclusion Criteria:

* Frozen sperm
* Frozen Embryo transfer
* Fresh cleavage stage embryo transfer
* Vanishing Twin Syndrome
* Fetal Reduction
* Preimlantation genetically screened embryo transfer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases undergoing ICSI in Ganin Fertility Center
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Gender ratio | 36-40 weeks after ICSI
  Neonatal gender ratio

CONTACTS AND LOCATIONS:
Overall Officials: khaled Elqusi, BSc, Principal Investigator — Ganin Fertility Center; Eman Hassanen, Bsc, Principal Investigator — Ganin Fertility Center; Hanaa Alkhader, ABB( ELD), Principal Investigator — Ganin Fertility Center; Hosam Zaki, MSc, FRCOG, Principal Investigator — Ganin Fertility Center; Ralph Henkel, PhD, Study Director — University of the Western Cape; Ashok Agarwal, PhD, Study Chair — American Center of Reproductive Medicine, Cleveland Clinic
Locations (1):
- Ganin Fertility Center, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Celik-Ozenci C, Jakab A, Kovacs T, Catalanotti J, Demir R, Bray-Ward P, Ward D, Huszar G. Sperm selection for ICSI: shape properties do not predict the absence or presence of numerical chromosomal aberrations. Hum Reprod. 2004 Sep;19(9):2052-9. doi: 10.1093/humrep/deh361. Epub 2004 Jun 17. PMID 15205404
- [Background] Avendano C, Franchi A, Taylor S, Morshedi M, Bocca S, Oehninger S. Fragmentation of DNA in morphologically normal human spermatozoa. Fertil Steril. 2009 Apr;91(4):1077-84. doi: 10.1016/j.fertnstert.2008.01.015. Epub 2008 Apr 28. PMID 18440529
- [Background] Said TM, Land JA. Effects of advanced selection methods on sperm quality and ART outcome: a systematic review. Hum Reprod Update. 2011 Nov-Dec;17(6):719-33. doi: 10.1093/humupd/dmr032. Epub 2011 Aug 25. PMID 21873262
- [Background] McElreavey K, Krausz C. Sex Chromosome Genetics '99. Male infertility and the Y chromosome. Am J Hum Genet. 1999 Apr;64(4):928-33. doi: 10.1086/302351. No abstract available. PMID 10090876
- [Background] Niederberger C. Absence of de novo Y-chromosome microdeletions in male children conceived through intracytoplasmic sperm injection. J Urol. 2005 Sep;174(3):1046. doi: 10.1097/01.ju.0000171902.28215.84. No abstract available. PMID 16094051
- [Background] Komori S, Kato H, Kobayashi S, Koyama K, Isojima S. Transmission of Y chromosomal microdeletions from father to son through intracytoplasmic sperm injection. J Hum Genet. 2002;47(9):465-8. doi: 10.1007/s100380200066. PMID 12202984
- [Result] Palermo G, Joris H, Devroey P, Van Steirteghem AC. Pregnancies after intracytoplasmic injection of single spermatozoon into an oocyte. Lancet. 1992 Jul 4;340(8810):17-8. doi: 10.1016/0140-6736(92)92425-f. PMID 1351601